CLINICAL TRIAL: NCT03957343
Title: Efficacy of the Pacing and Planning App for Persons With Mild Acquired Brain Injury
Brief Title: The Parkwood Pacing and Planning™ App
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: St. Joseph's Health Care (SJHC) Foundation (Unknown); Cowan Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 113428
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Acquired Brain Injury
Keywords: acquired brain injury; concussion
MeSH Terms: conditions — Brain Injuries; Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pacing and Planning App (Experimental): The Pacing and Planning Program is a points system to aid individuals with an acquired brain injury/concussion in planning daily activities and managing symptoms. Activities are allotted various points, depending on the energy the task requires and the symptoms they create. Activities can include anything from grocery shopping to driving or watching TV, etc. Patients are allotted a number of points for a day, and therefore learn to sparingly perform activities. This results in a reduction of symptoms and improved recovery time.
  Interventions: Device: Pacing and Planning App

INTERVENTIONS:
Device: Pacing and Planning App — Participants will download and use the Pacing and Planning app through mybrainpacer.ca. The app will be used to track and monitor their daily tasks and symptoms at any time, for as long as they would like to use the app. While using the app, participants will also fill out short assessments, including the Rivermead Post-Concussion Questionnaire once a month (to monitor symptoms) and an overall symptom question once a week (to rate how they feeling in general from a lot better to a lot worse).

SUMMARY:
In efforts to assist people who have had a concussion (mild traumatic brain injury), the Parkwood Pacing and Planning™ app has been developed and tested and will be released to the public. The app uses a point system where users have a daily point maximum assigned based on symptom severity with daily activities (recorded by the users). Users can then schedule their daily activities based on their allowed points. The goal is to help users with symptom self-management by facilitating activity planning and pacing.

Patients and clinicians have provided positive feedback on the initial version of the app. Using this as a foundation, the investigators envision enhancing the app to provide a more personalized user experience and to enable further discovery and innovations in the recovery from concussion. This will be accomplished through data analytics and machine-learning techniques, informed by the results of a large-scale research trial. This strategy will be used to customize the point system to facilitate the user with pacing and planning.

DETAILED DESCRIPTION:
At Parkwood Institute, the Outpatient Acquired Brain Injury Program receives approximately 350 referrals per year related to concussion (an increase of 500% since 2010). This program is renowned for its innovative programming, strong ties to brain injury research across the province, and the way that patients are engaged in program design, development and evaluation.

People who experience persistent and disabling problems three months beyond their brain injury are characterized as having "post-concussion syndrome". The list of post-concussion symptoms is long. Some of the most prevalent and debilitating symptoms include severe headaches and fatigue, forgetfulness, blurred vision and dizziness resulting in balance difficulties, poor concentration, sleep disturbances and depression. These symptoms can impact someone's daily functional ability, cause emotional distress and potentially limit their ability to return to work or school, which includes early back to work employment. Further, the impact of these debilitating symptoms can result in the breakdown of the family unit; whereby the patient's recovery is put at risk along with the mental health and financial impact on their family.

While trying to cope with these persistent symptoms, many individuals also experience a lack of post-recovery education and ongoing daily support as to how best to manage their symptoms while they begin to recover. Resting can actually prolong symptoms and lead to more difficulties, while being too active can restart or increase the severity of symptoms. However, health care providers at Parkwood Institute have discovered that patients who learn how to appropriately pace and plan their activities can minimize their symptoms, enhance recovery, and resume activities that had previously been a major part of their lives.

In 2013, the Parkwood Institute Outpatient Acquired Brain Injury Team developed a paper-based pacing and planning points system with a scale for rating the difficulty of daily activities (like grocery shopping, driving, and reading) according to the amount of energy each requires, and the severity of symptoms they trigger.

By tracking the maximum number of points they can comfortably expend in a day, patients learned how to self-manage their symptoms and improve participation in daily activities. In using this system, patients found they were able to reduce the severity and frequency with which symptoms occurred. A former outpatient said, "the points plan was such an effective way for me to get through the day without being utterly exhausted. I continue to use it as it has made me more independent, and as such, less reliant on my support people." In efforts to make this system more user-friendly and readily available for more patients, the investigators have created a mobile version of this planning and pacing points system, "MyBrainPacer™". Preliminary usability testing has indicated user and clinician satisfaction with the app.

For this next stage of development, the investigators plan to conduct a large-scale evaluation trial to demonstrate the effectiveness of the app more fulsomely. Completing this process will not only provide evidence related to the effectiveness of the app, but will also generate data to inform an existing gap in scientific literature: understanding of concussion recovery patterns. Analysis of the data will facilitate a better understanding of the patterns that exist between symptoms and everyday activity. In turn, this will enable development of a more personalized and customized version of the app, where the app 'learns' the patterns of a particular person and tailors their point system to their specific needs.

ELIGIBILITY:
Inclusion Criteria:

1. Experienced a mild traumatic brain injury/concussion
2. Disclosure of mechanism of injury and whether they were diagnosed with a mild traumatic brain injury/concussion by a registered health care practitioner
3. 18 yeas of age or older
4. Access to a smartphone or tablet
5. Able to read, write, and understand English

Exclusion Criteria:

1. Did not experience a mild traumatic brain injury/concussion
2. Unwilling to disclose mechanism of injury and whether they were diagnosed with a mild traumatic brain injury/concussion
3. Under 18 years of age
4. No access to a smartphone or tablet
5. Inability to read, write, and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Symptom changes | Approximately 3 years
  These are assessed using the Rivermead Post Concussion Questionnaire (RPQ). The RPQ evaluates the severity of 16 common post-concussion symptoms over the past 24 hours (e.g. headache, sleep disturbance, and noise sensitivity). It is a 5-point scale from 0-4, where 0 indicates no symptoms (better outcome), and 4 indicates the symptom is a severe problem (worse outcome). The total from each symptom can be summed for a total score out of 64, where 64 represents experiencing all symptoms, and they are all a severe problem (worse outcome). This will contribute to understanding the effectiveness of the app.
Changes in general well-being | Approximately 3 years
  This will be assessed using the responses to one bi-weekly question. The bi-weekly question asks how users are feeling, and they can choose to answer with much worse, worse, the same, better, or much better. This will contribute to understanding the effectiveness of the app.

SECONDARY OUTCOMES:
Change in daily activities and symptoms | Approximately 3 years
  This will be measured through reported activities and symptoms. Participants will be able to input the activities (e.g. reading), the time spent doing that activity (e.g. 20 minutes) and their points and difficulty associated with the activity (maximum 10, where 0 is no difficulty and not experiencing symptoms and 10 is extremely difficult and experiencing symptoms). Accordingly, this data will be used to determine recovery patterns and increase personalization of the app.

CONTACTS AND LOCATIONS:
Overall Officials: Dalton Wolfe, PhD, Principal Investigator — Lawson Health Research Institiute
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers.

REFERENCES:
- [Background] Savola O, Hillbom M. Early predictors of post-concussion symptoms in patients with mild head injury. Eur J Neurol. 2003 Mar;10(2):175-81. doi: 10.1046/j.1468-1331.2003.00552.x. PMID 12603294
- [Background] Schneider KJ, Leddy JJ, Guskiewicz KM, Seifert T, McCrea M, Silverberg ND, Feddermann-Demont N, Iverson GL, Hayden A, Makdissi M. Rest and treatment/rehabilitation following sport-related concussion: a systematic review. Br J Sports Med. 2017 Jun;51(12):930-934. doi: 10.1136/bjsports-2016-097475. Epub 2017 Mar 24. PMID 28341726